CLINICAL TRIAL: NCT02280187
Title: InductOs® in Real World Spine Surgery; A Retrospective, French, Multi-centric, Study
Acronym: InductOR
Status: Completed | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2.05.8005
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Spine Fusion
Keywords: InductOs; rhBMP-2; Retrospective; France; Fusion; real world use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spine Fusion with InductOs: Patient had spinal fusion surgery with InductOs between 1st January 2011 and 31st December 2012
  Interventions: Procedure: Spine Fusion

INTERVENTIONS:
Procedure: Spine Fusion — All patients have been treated with a spinal fusion procedure with InductOs (rhBMP-2/ACS) following standard practice in each center.

SUMMARY:
It is a phase IV, national, multicenter, observational, retrospective study collecting data from patient medical files in French spinal centers.

The aim of the study is to describe the real world use of InductOs in Spine fusion in France.

Approximately 10 French centers will enroll 400 patients. The retrospective review of records will focus on patients who have undergone a spinal fusion surgery. Patient should be considered for enrollment if he/she has been treated with InductOs between January 1, 2011 and 31st December 2012.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has had spinal fusion surgery with InductOs between 1st January 2011 and 31st December 2012
2. Patient as medical records documenting Study Procedure with at least: Age, sex, medical history, primary diagnostic indication, level(s) treated, procedure(s) type, interbody device's information if used
3. Patient has received the "information and non-objection letter" and reception is confirmed by registered courier
4. Patient is ≥18 years old at the date of the Study Procedure

Exclusion Criteria:

1. Patient declines participation
2. Vulnerable patients, unable to understand the non-objection letter or unable to exercise free decision to refuse to participate to the study (at investigator's discretion)
3. Patient died since study procedure*
4. Participation in concurrent interventional trial during study participation (from Study Procedure to last study follow-up) which may confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The retrospective review of records will focus on patients who have undergone a spinal fusion surgery. Patient should be considered for enrollment if he/she has been treated with InductOs between January 1, 2011 and 31st December 2012.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Passuti, Pr, Principal Investigator — Nantes University Hospital
Locations (10):
- France (10):
  - CHU de Bordeaux- Centre Universitaire Pellegrin, Bordeaux
  - Centre Orthopedique Santy, Lyon
  - Hopital De La Timone Adultes, Marseille
  - Hopital Prive Clairval, Marseille
  - CHU de Nantes, Nantes
  - Centre Hospitalier Universitaire Nice - Hôpital Pasteur, Nice
  - Nouvelle Clinique De L'Union, Saint-Jean
  - Clinique Du Parc à Saint -Priest en Jarez, Saint-Priest-en-Jarez
  - Hopital Civil, Strasbourg
  - Clinique Medipole Garonne, Toulouse

RESULTS

PARTICIPANT FLOW:
Groups:
- Spine Fusion With InductOs: Patient has had spinal fusion surgery with InductOs between 1st January 2011 and 31st December 2012
  Spine Fusion: All patients have been treated with a spinal fusion procedure with InductOs (rhBMP-2/ACS) following standard practice in each center.
Period: Overall Study
Arm/Group | Spine Fusion With InductOs
Started | 400
Completed | 182
Not Completed | 218
Not completed — Lost to Follow-up | 218

BASELINE CHARACTERISTICS:
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (14.8)
Gender [Count of Participants; unit: Participants]
  Female | 237
  Male | 163
Smoking Status [Number; unit: participants]
  Current smoker | 110
  Not currently smoking | 267
  Not available | 23
Medical history with or without Diabetes [Number; unit: participants]
  Diabetics | 29
  Non-diabetics | 371

OUTCOME MEASURES:

1. Primary Outcome: The Primary Diagnostic Indication for InductOs Use
Description: The primary diagnostic indications, which patients were treated with InductOs during spine fusion surgery in France, are presented.
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
percentage of participants
  Degenerative disc disease (DDD) | 32.3
  Disc herniation | 4.5
  Stenosis | 3.5
  Spondylolisthesis | 29.8
  Spondylosis (e.g. osteoarthritis) | 0.8
  Deformity (i.e. Scoliosis, kyphosis) | 14.8
  Pseudoarthrosis | 7.3
  Trauma | 2.3
  Other | 5.0

2. Primary Outcome: Spine Levels Treated
Description: The number of spine levels from the occiput to S1 is presented.
Time Frame: During surgery
Measure: Number; unit: spine level
Units Other Than Participants: Spine level
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
Number analyzed (Spine level) | 634
spine level
  Occiput-C1 | 0
  C1-C2 | 1
  C2-C3 | 0
  C3-C4 | 0
  C4-C5 | 0
  C5-C6 | 0
  C6-C7 | 0
  C7-T1 | 0
  T1-T2 | 0
  T2-T3 | 2
  T3-T4 | 2
  T4-T5 | 3
  T5-T6 | 4
  T6-T7 | 5
  T7-T8 | 3
  T8-T9 | 4
  T9-T10 | 5
  T10-T11 | 8
  T11-T12 | 9
  T12-L1 | 15
  L1-L2 | 18
  L2-L3 | 46
  L3-L4 | 106
  L4-L5 | 214
  L5-S1 | 189

3. Primary Outcome: Primary Surgical Approaches Used for Implantation of InductOs
Description: The surgical approaches for implanting InductOs are classified as anterior lumbar interbody fusion (ALIF), posterior lumbar interbody fusion (PLIF), translateral lumbar interbody fusion (TLIF), lateral lumber interbody fusion (LLIF, including DLIF and XLIF), posterolateral fusion (PLF). The number of spine levels by surgical approaches is presented.
Time Frame: During surgery
Measure: Number; unit: spine level
Units Other Than Participants: Spine level
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
Number analyzed (Spine level) | 634
spine level
  ALIF | 188
  PLIF | 111
  TLIF | 4
  LLIF | 106
  PLF | 221
  Other | 4

4. Primary Outcome: The Interbody Device Brand/Generic Names Used With InductOs
Description: The number of spine levels with InductOs is presented by interbody brand/generic names.
Time Frame: during surgery
Measure: Number; unit: spine level
Units Other Than Participants: Spine level
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
Number analyzed (Spine level) | 634
spine level
  Capstone | 26
  Crescent | 3
  Juliet An | 2
  Perimeter | 91
  Pyramesh | 4
  Roi | 43
  Roi-A | 26
  Roi-T | 5
  Sovereign | 45
  Synfix-Lr | 9
  Vlift | 5
  Other | 96
  No Cage Used | 271
  Not Available | 8

5. Primary Outcome: Placement of the Matrix Wetted With InductOs
Description: The placement of the matrix was classified as posterior lateral or interbody space (Inside the cage, between the cages or outside the cage) or any other placement specified. The number of spine levels is presented by placement of the matrix.
Time Frame: During surgery
Population: The total levels across all the rows are higher than total number of levels analyzed because multiple answers are possible.
Measure: Number; unit: spine level
Units Other Than Participants: Spine level
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
Number analyzed (Spine level) | 634
spine level
  Posterior lateral | 270
  Interbody (inside the cage) | 335
  Interbody (between the cage) | 60
  Interbody (outside cage) | 22
  Other placement | 20

6. Primary Outcome: Supplemental Fixation
Description: The number of spine levels on which supplemental fixation was performed is presented by approaches of stabilization (anterior or posterior stabilization).
Time Frame: During surgery
Population: The total levels across all the rows are higher than total number of levels analyzed because some levels may be represented in more than one rows.
Measure: Number; unit: spine level
Units Other Than Participants: Spine level
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
Number analyzed (Spine level) | 634
spine level
  Anterior stabilization | 200
  Posterior stabilization | 399
  No stabilization | 99

7. Primary Outcome: Instrumentations Used for Stabilization
Description: The number of spine levels using instrumentations for stabilization is presented by types of instrumentations.
Time Frame: during surgery
Population: The total levels in the summary are higher than total amount of levels because multiple answers are possible.
Measure: Number; unit: spine level
Units Other Than Participants: Spine level
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
Number analyzed (Spine level) | 634
spine level
  Screws | 454
  Rods | 394
  Plates | 105
  Other | 77

8. Secondary Outcome: The Number of Adverse Events of Interest
Description: An adverse event was considered an event of interest (AEI) if an adverse event was considered important to follow. These included reactions described in the EU product label, events monitored in the EU Risk Management Plan, events that were considered possible related to the treatment by the investigator, and events that had serious health consequences for patients (e.g. hospitalization).
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
events | 31

9. Secondary Outcome: AEI Categorisation
Description: The number of AEIs is presented by the categories predefined in the study protocol. The AEI MedDRA coded terms are presented in Section of serious adverse event.
Time Frame: 12 months
Measure: Number; unit: events
Units Other Than Participants: adverse event
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
Number analyzed (adverse event) | 31
events
  Exuberant bone formation/heterotopic bone growth | 0
  Excessive bone resorption | 1
  Nerve compression or nerve root disorders | 3
  Allergic reactions or inflammation | 1
  Fluid collection at the site of implant | 5
  Device (implant) displacement | 7
  Male fertility problems | 1
  Neoplasms (benign, malignant,and unspecified) | 1
  Other Adverse Event of interest | 12

10. Secondary Outcome: The Number of Subjects Having Secondary Spine Surgical Intervention
Description: The number of subjects who had secondary spine surgical intervention at index level treated with InductOs and other level (either never treated or treated without InductOs) through 12 months is reported.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
participants
  subjects having planned secondary spine surgery | 3
  subjects having unplanned secondary spine surgery | 9

11. Secondary Outcome: The Number of Unplanned Secondary Spine Interventions in Subgroups
Description: The number of unplanned secondary spine interventions is reported by subgroups (smoker, non-smoker, diabetics, and non-diabetics).
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 400
participants
  unplanned secondary surgeries in smokers (n=110) | 2
  unplanned secondary surgeries in nonsmokers(n=267) | 1
  unplanned secondary surgeries-diabetics (n=29) | 0
  unplanned secondary surgeries-nondiabetics (n=371) | 3

12. Secondary Outcome: Fusion Status at the Last Assessment Performed by 12 Months
Description: According to the study protocol, fusion status was determined to be either success or no success based on the images. If fusion failed at 1 level, the fusion was considered to be failed for the patient. The fusion rate at the last assessment is reported.
Time Frame: 12 months
Population: The subjects with the image that unable to determine fusion status and the assessment not done" were not taken into account.
Measure: Number; unit: percentage of participants
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 266
percentage of participants
  Fusion success | 73.3
  Fusion failed | 26.7

13. Secondary Outcome: Fusion Rates in Subgroups
Description: Fusion rates in subgroup (Smokers, non-smokers, Patients with and without diabetes) are reported.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Spine Fusion With InductOs
Number analyzed (Participants) | 266
percentage of participants
  Successful fusion rate in smokers (n=77) | 72.7
  Successful fusion rate in non-smokers (n=179) | 74.3
  Successful fusion rate in diabetics (n=14) | 78.6
  Successful fusion rate in non-diabetics (n=252) | 73.0

ADVERSE EVENTS:
Time Frame: 12 months
Description: This is a retrospective study. During this study, all Adverse Events of Interest (AEIs) that occurred after the application of InductOs were collected. Please see secondary outcome 8 (the number of AEIs) for the definition of AEI. The table below contains all AEI, regardless of seriousness.
Arm/Group | Spine Fusion With InductOs
Serious Adverse Events (participants affected / at risk) | 27/400
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spine Fusion With InductOs (N=400)
Meningocele (Congenital, familial and genetic disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Device Breakage (General disorders) | 1 (1)
Device Deployment Issue (General disorders) | 1 (1)
Device Dislocation (General disorders) | 2 (2)
Implant Site Haematoma (General disorders) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 1 (1)
Endocarditis Staphylococcal (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Wound Infection Staphylococcal (Infections and infestations) | 1 (1)
Extradural Haematoma (Injury, poisoning and procedural complications) | 2 (2)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 2 (2)
Post Procedural Inflammation (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Spinal Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1)
Motor Dysfunction (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Radiculitis Lumbosacral (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Spinal Cord Ischaemia (Nervous system disorders) | 1 (1)
Retrograde Ejaculation (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less